CLINICAL TRIAL: NCT02598310
Title: Phase II Study of Neoadjuvant Nab-paclitaxel (PTX) and Trastuzumab for ER Negative and HER2 Positive Breast Cancer
Brief Title: Neoadjuvant Nab-PTX and Trastuzumab for ER Negative and HER2 Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Osaka Medical College (Other)
Responsible Party: Principal Investigator, Satoru Tanaka, MD, PhD, Osaka Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMC BC-04; OMC BC-04 (Other: Osaka Medical College)
Record Dates: First submitted 2015-11-02; First posted 2015-11-05 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Estrogen Receptor Negative Neoplasm; HER-2 Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nab-paclitaxel plus trastuzumab (Experimental): Four cycles of nab-PTX 260 mg/m2 with trastuzumab 6 mg/kg (8 mg/kg as the loading dose). One year of adjuvant trastuzumab will be administrated. Anthracycline regimens may be administered by physician's choice for the case expected to have a high risk of recurrence based on the pathological findings of surgical specimen. Adjuvant endocrine therapy may be administrated for the case with weakly hormone-sensitive (1-9% of positive cells) tumor.
  Interventions: Drug: nab-paclitaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: nab-paclitaxel — nab-paclitaxel 260mg/m2 q3w
  Other Names: Abraxane
Drug: Trastuzumab — trastuzumab 6 mg/kg (8 mg/kg as the loading dose)
  Other Names: Herceptin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of nab-PTX and trastuzumab for ER negative and HER2 positive operable (tumor size of 3cm or less and N0) breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive breast cancer
2. Tumor size of 3cm or less and N0
3. Hormone receptors have been identified as negative
4. HER2 positive confirmed by IHC 3+ or FISH+
5. LVEF > 50% by echocardiogram or MUGA
6. Adequate EKG
7. No prior treatment for breast cancer
8. PS 0-1
9. Required baseline laboratory data WBC > 4,000/mm3 and Neut > 2,000/mm3 PLT > 100,000/mm3 Hb > 9.0g/dl AST and ALT < ULNx2.5 T-Bil < 1.5mg/dl Serum creatinin < 1.5mg/dl
10. Written informed consent

Exclusion Criteria:

1. With history of hypersensitivity reaction for important drug in this study
2. With history of invasive breast cancer
3. Bilateral invasive breast cancer
4. Patients with medical conditions that renders them intolerant to primary chemotherapy and related treatment, including infection, diarrhea, intestinal paralysis, severe Diabetes Mellitus
5. Positive for HBs antigen or HCV antibody
6. With history of congestive heart failure, uncontrolled or symptomatic angina pectoris, arrhythmia or myocardial infarction, poorly controlled hypertension
7. With severe edema
8. With severe peripheral neuropathy
9. With severe psychiatric disorder
10. Pregnant or nursing women
11. The case that is judged to be unsuitable for this study by physician

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Pathological complete response rate | Up to 12 weeks after the protocol therapy

SECONDARY OUTCOMES:
Disease free survival | Five years after the last patient enrolled
Objective response rate | Up to 6 weeks after the protocol therapy
Pathological response rate | Up to 12 weeks after the protocol therapy
Breast-conserving surgery rate | Up to 6 weeks after the protocol therapy
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 6 weeks after the protocol therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuhiko Iwamoto, MD, PhD, Principal Investigator — Osaka Medical College
Locations (1):
- Osaka Medical College, Takatsuki, Osaka, Japan

REFERENCES:
- [Derived] Tanaka S, Matsunami N, Morishima H, Oda N, Takashima T, Noda S, Kashiwagi S, Tauchi Y, Asano Y, Kimura K, Fujioka H, Terasawa R, Kawaguchi K, Ikari A, Morimoto T, Michishita S, Kobayashi T, Sakane J, Nitta T, Sato N, Hokimoto N, Nishida Y, Iwamoto M. De-escalated neoadjuvant therapy with nanoparticle albumin-bound paclitaxel and trastuzumab for low-risk pure HER2 breast cancer. Cancer Chemother Pharmacol. 2019 Jun;83(6):1099-1104. doi: 10.1007/s00280-019-03836-z. Epub 2019 Apr 8. PMID 30963212